CLINICAL TRIAL: NCT01518608
Title: Alfentanil and the Elimination of Sympathetic Responses to Tracheal Intubation During Rapid Sequence Induction of Anesthesia: A Probability-based Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Aker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29237403/SMR-1651
Record Dates: First submitted 2011-08-25; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia Intubation Complication
Keywords: Alfentanil; Tracheal intubation; Rapid sequence induction
MeSH Terms: interventions — Alfentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfentanil 0.5mg/ml (Rapifen , Janssen-Cilag) — Induction dose(0µg/kg,10µg/kg,20µg/kg,30µg/kg,40µg/kg,50µg/Kg,and 60µg/kg) 12 patients in each dose group.
  Pentothal 4mg/kg Rocuronium 0.6 mg/kg

SUMMARY:
Induction of anesthesia:

After 3 minutes pre-oxygenation with 100% oxygen, a blinded dose alfentanil (0,10,20,30,40,50 or 60 µg/kg, followed by thiopental 4 mg/kg and rocuronium 0.6 mg/kg will be administered over 15 sec. Laryngoscopy will be performed 40 s. after injection of rocuronium, with the goal being to have the endotracheal tube passed through the patients vocal cords and the cuff inflated within the following 15 s . The investigator performing the tracheal intubation is blinded to the dose of alfentanil administered.

Blood samples:

As part of the study efficacy, blood samples, will be collected prior to induction and 30 s., 1 min. 3 min. and 5 min postintubation to determine blood concentrations of alfentanil and catecholamines.

DETAILED DESCRIPTION:
Introduction:

Autonomic responses (blood pressure and heart rate increases) secondary to tracheal intubation are probably not harmful to healthy individuals(1). However, in certain groups of patients (cardiac/neurosurgical/ophthalmic surgery), strict control of these responses during anesthesia may add to the safety of patient care (2-6).

Traditionally, rapid sequence induction (RSI) of anesthesia is performed with combined administration of pentothal and suxamethonium. Significant increases in blood pressure and heart rate will be observed in most patients when this drug regimen is used(7-9). Opioid drugs may obtund autonomic responses to tracheal stimulation(10), but at present there is no consensus regarding the use of opioids as an integral part of the RSI of anesthesia.

AIMS & OBJECTIVES:

* Define guidelines for proper care of cardiac/neurosurgical/eye surgery patients during induction of anesthesia when rapid airway control is needed.
* Determine the dose of alfentanil needed to prevent blood pressure and heart rate increases > 10% secondary to tracheal intubation performed in a rapid-sequence fashion (intubation completed within 70 s after start of drug administration: alfentanil-pentothal 4 mg/kg-rocuronium 0.6 mg/kg).
* Determine the optimal dose of alfentanil to obtain perfect conditions for tracheal intubation in healthy surgical patients when laryngoscopy is initiated within 55 s after start of drug administration (alfentanil-pentothal 4 mg/kg-rocuronium 0,6 mg/kg).

Induction of anesthesia:

After 3 min pre-oxygenation with 100% oxygen, a blinded dose of alfentanil (0, 10, 20, 30, 40, 50 or 60 mcg/kg), followed by thiopental 4 mg/kg and rocuronium 0.6 mg/kg will be administered over 15 s. Cricoid pressure will be applied when the patient is unconscious.

Laryngoscopy and intubation:

Laryngoscopy will be performed 40 s after injection of rocuronium, with the goal being to have the endotracheal tube passed through the patients vocal cords and the cuff inflated within the following 15 s. The investigator performing the tracheal intubation will be blinded to the dose of alfentanil administered.

Maintenance of anesthesia:

The study ends 5 min post intubation. At this time sevoflurane and fentanyl will be administered according to the patient's needs. Ventilation will be adjusted to pCO2-values in the range 4.5-6 kPa, and body temperature maintained at > 36 degree ºC with a forced-air warmer.

Monitoring:

Routine monitoring of blood pressure, ECG, and pulse oximetry, according to standard of anaesthesia, approved by the Society of the Norwegian Anaesthesiologists. An arterial line will be inserted in one of the radial arteries for accurate beat-to-beat recording of blood pressure and heart rate, and for collection of blood samples.

Statistical analysis plan:

In the present study a nonlinear logistic regression analysis will be used to determine the optimal dose of alfentanil based on the success rates of optimal blood pressure control (blood pressure increase < 10%)and the success rates of perfect intubation conditions in all alfentanil dose groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients and admitted for elective surgery.
* Aged 18-55 years
* Written informed consent

Exclusion Criteria:

* Body Mass Index (BMI) > 28 Kg/m²
* Patients with known allergy to study drug
* Patients with known porphyria
* Neuromuscular disease or undergoing treatment with drugs known to interfere with neuromuscular transmission.
* Mallampati class > 2airway anatomy, or anticipated difficulty with mask ventilation or tracheal intubation.
* Neuromuscular disease
* Pulmonary disease
* Cardiovascular disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Alfentanil and blockage of sympathetic responses: A dose-response study. | 2 years
  Effectivness of controling Blood pressure during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Tom Heier, MD, Phd., Study Director — University of Oslo
Locations (2):
- Norway (2):
  - Oslo University Hospital/ Aker, Oslo, Akershus
  - Oslo University Hospital / Aker, Oslo

REFERENCES:
- [Derived] Abou-Arab MH, Feiner JR, Spigset O, Heier T. Alfentanil during rapid sequence induction with thiopental 4 mg/kg and rocuronium 0.6 mg/kg: tracheal intubation conditions. Acta Anaesthesiol Scand. 2015 Nov;59(10):1278-86. doi: 10.1111/aas.12584. Epub 2015 Jul 14. PMID 26176994